CLINICAL TRIAL: NCT01079780
Title: A Randomized Phase II Study of Irinotecan and Cetuximab With or Without the Anti-Angiogenic Antibody, Ramucirumab (IMC-1121B), in Advanced, K-ras Wild-Type Colorectal Cancer Following Progression on Bevacizumab-Containing Chemotherapy
Brief Title: Irinotecan Hydrochloride and Cetuximab With or Without Ramucirumab in Treating Patients With Advanced Colorectal Cancer With Progressive Disease After Treatment With Bevacizumab-Containing Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7208; CDR0000666736
Record Dates: First submitted 2010-03-02; First posted 2010-03-03 (Estimated); Results first posted 2022-06-10 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Colorectal Cancer
Keywords: mucinous adenocarcinoma of the colon; recurrent colon cancer; signet ring adenocarcinoma of the colon; stage III colon cancer; stage IV colon cancer; mucinous adenocarcinoma of the rectum; recurrent rectal cancer; signet ring adenocarcinoma of the rectum; stage III rectal cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Cetuximab; Ramucirumab; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (IC) (Active Comparator): Patients receive cetuximab (500 mg/m2) intravenously (IV) over 60-120 minutes and irinotecan hydrochloride (180 mg/m2) over 60-90 minutes on day 1. Treatment repeats every 2 weeks until disease progression or unacceptable toxicities.
  Interventions: Biological: cetuximab; Drug: irinotecan hydrochloride
- Arm B (ICR) (Experimental): Patients receive ramucirumab (8 mg/kg) IV over 60 minutes on day 1 and cetuximab and irinotecan hydrochloride as in arm A. Treatment repeats every 2 weeks until disease progression or unacceptable toxicities.
  Interventions: Biological: cetuximab; Biological: ramucirumab; Drug: irinotecan hydrochloride
- Arm C (mICR) (Experimental): Patients receive reduced dose of ramucirumab (6 mg/kg) IV over 60 minutes on day 1 and cetuximab (150 mg/m2) and irinotecan hydrochloride (400 mg/m2) as in arm B. Treatment repeats every 2 weeks until disease progression or unacceptable toxicities.
  Interventions: Biological: cetuximab; Biological: ramucirumab; Drug: irinotecan hydrochloride

INTERVENTIONS:
Biological: cetuximab — Given IV
  Other Names: IMC-C225; Erbitux®; NSC-714692
Biological: ramucirumab — Given IV
  Other Names: IMC 1121B; 1121B
  Arms: Arm B (ICR); Arm C (mICR)
Drug: irinotecan hydrochloride — Given IV
  Other Names: Irinotecan hydrochloride trihydrate

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as irinotecan hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as cetuximab and ramucirumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Cetuximab and ramucirumab may also stop the growth of colorectal cancer by blocking blood flow to the tumor. It is not yet know whether giving cetuximab and irinotecan hydrochloride together is more effective with or without ramucirumab in treating colorectal cancer.

PURPOSE: This randomized phase II trial is studying the side effects and how well giving cetuximab and irinotecan hydrochloride with or without ramucirumab work in treating patients with advanced colorectal cancer with progressive disease after treatment with bevacizumab-containing chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate the progression-free survival of patients with advanced K-ras wild-type colorectal cancer, following progression on bevacizumab-contained chemotherapy, treated with irinotecan hydrochloride and cetuximab with versus without ramucirumab as second-line therapy.
* To evaluate the response rate in patients treated with these regimens.
* To evaluate the grade 3-4 toxicity rates of these regimens in these patients.
* To evaluate the overall survival of patients treated with these regimens.

OUTLINE: This is a multicenter, randomized study. Patients are stratified according to performance status (0 vs 1), discontinuation of oxaliplatin before disease progression (yes vs no), and time to disease progression since last treatment (≤ 6 months vs > 6 months). Patients are randomized to 1 of 2 treatment arms.

* Arm A: Patients receive cetuximab IV over 60-120 minutes and irinotecan hydrochloride over 60-90 minutes on day 1.
* Arm B: Patients receive ramucirumab IV over 60 minutes on day 1 and cetuximab and irinotecan hydrochloride as in arm A. Arm B was closed early due to excessive toxicities and Arm C was then added to the study with reduced dose of protocol drugs.
* Arm C: Patients receive reduced dose of ramucirumab, cetuximab and irinotecan hydrochloride as in arm B.

In all arms, courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up periodically for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Measurable disease
* Histologically confirmed adenocarcinoma of the colon or rectum
* K-ras wild type based on either primary or metastatic tumor
* Must have received prior first-line therapy comprising oxaliplatin-based fluoropyrimidine-containing chemotherapy and bevacizumab for metastatic colorectal cancer
* Registration within 42 days since confirmed disease progression
* Performance status 0-1
* ANC ≥ 1,500/μL
* Platelet count ≥ 75,000/μL
* Hemoglobin ≥ 9 g/dL
* Serum creatinine ≤ 1.5 times upper limit of normal (ULN) OR creatinine clearance ≥ 40 mL/min
* Urine protein ≤ 1+ on dipstick or routine urinalysis (if ≥ 2+, a 24-hour urine collection must demonstrate < 1,000 mg of protein)
* Total bilirubin ≤ 2.0 mg/dL
* AST and ALT ≤ 3.0 times ULN (5.0 times ULN for patients with liver metastases)
* INR ≤ 1.6 (≤ 3.0 for patients on warfarin and no active bleeding [i.e., no bleeding within the past 14 days])
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study therapy
* At least 28 days and no more than 90 days since prior bevacizumab
* Concurrent stable dose of oral anticoagulant or low-molecular weight heparin allowed

Exclusion Criteria:

* Brain or CNS metastases
* Pregnant or nursing
* Prior therapy with drugs other than oxaliplatin and a fluoropyrimidine plus bevacizumab for colorectal cancer
* Clinically significant (equivalent to NCI CTCAE grade 3-4) bleeding episodes within the past 3 months
* Active infection
* Symptomatic congestive heart failure
* Unstable angina pectoris
* Symptomatic or poorly controlled cardiac arrhythmia
* Uncontrolled thrombotic or hemorrhagic disorder
* Uncontrolled or poorly controlled hypertension despite standard medical management (e.g., consistently systolic BP > 160 mm Hg and diastolic BP > 90 mm Hg)
* Acute arterial thrombotic events within the past 6 months, including cerebrovascular accident, transient ischemic attack, myocardial infarction, or unstable angina
* Other cancer requiring therapy within the past 3 years except in situ carcinoma or nonmelanoma skin cancer
* Acute or subacute intestinal obstruction
* History of inflammatory bowel disease requiring pharmacological and/or surgical intervention within the past 12 months
* Known allergy to any of the treatment components
* Major surgery within the past 28 days
* Subcutaneous venous access device placement within the past 7 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2011-01-18 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2021-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard S. Hochster, MD, Principal Investigator — NYU Langone Health
Locations (255):
- United States (255):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Yale Cancer Center, New Haven, Connecticut
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Nancy N. and J. C. Lewis Cancer and Research Pavilion at St. Joseph's/Candler, Savannah, Georgia
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Kellogg Cancer Care Center, Highland Park, Illinois
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - Provena St. Mary's Regional Cancer Center - Kankakee, Kankakee, Illinois
  - North Shore Oncology and Hematology Associates, Limited - Libertyville, Libertyville, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Cancer Care and Hematology Specialists of Chicagoland - Niles, Niles, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - West Suburban Center for Cancer Care, River Forest, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - Hematology Oncology Associates - Skokie, Skokie, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - William N. Wishard Memorial Hospital, Indianapolis, Indiana
  - Clarian Arnett Cancer Care, Lafayette, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - McPherson, McPherson, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - Ochsner Health Center - Bluebonnet, Baton Rouge, Louisiana
  - Ochsner Health Center - Covington, Covington, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Medical Center of Louisiana - New Orleans, New Orleans, Louisiana
  - Ochsner Cancer Institute at Ochsner Clinic Foundation, New Orleans, Louisiana
  - Greater Baltimore Medical Center Cancer Center, Baltimore, Maryland
  - Baystate Regional Cancer Program at D'Amour Center for Cancer Care, Springfield, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology - Woodbury, Woodbury, Minnesota
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - Hunterdon Regional Cancer Center at Hunterdon Medical Center, Flemington, New Jersey
  - CentraState Medical Center, Freehold, New Jersey
  - Hematology Oncology Associates, PC, Albuquerque, New Mexico
  - Presbyterian Cancer Treatment Center at Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New Mexico Cancer Care Associates, Santa Fe, New Mexico
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - Roger Maris Cancer Center at MeritCare Hospital, Fargo, North Dakota
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Wood County Oncology Center, Bowling Green, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - MetroHealth Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Community Cancer Center, Elyria, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - St. Luke's Cancer Network at St. Luke's Hospital, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Doylestown Hospital Cancer Center, Doylestown, Pennsylvania
  - PinnacleHealth Regional Cancer Center at Polyclinic Hospital, Harrisburg, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Cancer Center of Paoli Memorial Hospital, Paoli, Pennsylvania
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Joan Karnell Cancer Center at Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - Pottstown Memorial Regional Cancer Center, Pottstown, Pennsylvania
  - McGlinn Family Regional Cancer Center at Reading Hospital and Medical Center, Reading, Pennsylvania
  - Hematology and Oncology Associates of Northeastern Pennsylvania, Scranton, Pennsylvania
  - Grand View Hospital, Sellersville, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - CCOP - Main Line Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Parkland Memorial Hospital, Dallas, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - West Virginia University Health Sciences Center - Charleston, Charleston, West Virginia
  - Langlade Memorial Hospital, Antigo, Wisconsin
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Vince Lombardi Cancer Clinic - Green Bay at Aurora BayCare Medical Center, Green Bay, Wisconsin
  - UW Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Vince Lombardi Cancer Clinic - Marinette, Marinette, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - Regional Cancer Center at Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - St. Nicholas Hospital, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic - Sheboygan, Sheboygan, Wisconsin
  - Marshfield Clinic at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Aurora Medical Center, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic - Two Rivers, Two Rivers, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin
  - University of Wisconcin Cancer Center at Aspirus Wausau Hospital, Wausau, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Riverview UW Cancer Center at Riverview Hospital, Wisconsin Rapids, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be made available upon request as per the ECOG-ACRIN Data Sharing Policy.

REFERENCES:
- [Derived] Hochster HS, Catalano P, Weitz M, Mitchell EP, Cohen D, O'Dwyer PJ, Faller BA, Kortmansky JS, O'Hara MH, Kricher SM, Lacy J, Lenz HJ, Verma U, Benson AB. Combining antivascular endothelial growth factor and anti-epidermal growth factor receptor antibodies: randomized phase II study of irinotecan and cetuximab with/without ramucirumab in second-line colorectal cancer (ECOG-ACRIN E7208). J Natl Cancer Inst. 2024 Sep 1;116(9):1487-1494. doi: 10.1093/jnci/djae114. PMID 38775718

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was accrued on January 18, 2011.
Groups:
- Arm A (IC): Patients receive cetuximab (500 mg/m^2) intravenously (IV) over 60-120 minutes and irinotecan hydrochloride (180 mg/m^2) over 60-90 minutes on day 1. Treatment repeats every 2 weeks until disease progression or unacceptable toxicities.
- Arm C (mICR): Patients receive reduced dose of ramucirumab (6 mg/kg) IV over 60 minutes on day 1 and cetuximab (150 mg/m^2) and irinotecan hydrochloride (400 mg/m^2) as in arm B. Treatment repeats every 2 weeks until disease progression or unacceptable toxicities.
Period: Overall Study
Arm/Group | Arm A (IC) | Arm B (ICR) | Arm C (mICR)
Started | 70 | 16 | 50
Started Protocol Therapy | 69 | 16 | 48
Treated Patients With Toxicity Data Available | 68 | 16 | 48
Eligible and Treated | 62 | 16 | 45
Analyzable Patients for Efficacy Analysis | 44 | 0 | 45
Completed | 0 | 0 | 0
Not Completed | 70 | 16 | 50
Not completed — Disease progression | 43 | 7 | 31
Not completed — Adverse Event | 13 | 5 | 7
Not completed — Death | 2 | 0 | 2
Not completed — Withdrawal by Subject | 6 | 4 | 4
Not completed — Alternative therapy | 2 | 0 | 2
Not completed — Physician Decision | 1 | 0 | 1
Not completed — Error made in lesion measurement | 1 | 0 | 0
Not completed — Patient had surgery | 1 | 0 | 0
Not completed — Treatment cycle delay | 0 | 0 | 1
Not completed — Never started treatment | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients are included in this analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (IC) | Arm B (ICR) | Arm C (mICR) | Total
Number analyzed (Participants) | 62 | 16 | 45 | 123
Age, Continuous [Median (Full Range); unit: years] | 59.8 [34 to 84] | 60.0 [43 to 76] | 60.4 [37 to 80] | 60.3 [34 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 7 | 13 | 45
  Male | 37 | 9 | 32 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 5 | 12
  Not Hispanic or Latino | 54 | 13 | 38 | 105
  Unknown or Not Reported | 3 | 1 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 12 | 1 | 3 | 16
  White | 47 | 15 | 37 | 99
  More than one race | 1 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-fee survival is defined as the time from randomization to disease progression or death without documentation of progression. Censoring occurred at the date of last disease assessment without progression for cases without documentation of progression, except for cases where death occurred within a short period of time (4 months) following the date last known progression-free, in which case the death was considered an event.
  Progression is defined as appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions or at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: Assessed every 3 months for 2 years, every 6 months for the 3rd year, then annually up to 5 years
Population: Only eligible patients are included in this analysis. For the comparison between arms A and C, only eligible patients that were concurrently randomized were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (IC) | Arm B (ICR) | Arm C (mICR)
Number analyzed (Participants) | 44 | 16 | 45
months | 5.98 [3.88 to 9.07] | 7.03 [3.91 to 10.32] | 9.20 [5.52 to 11.33]
Statistical Analysis 1: Comparison: Arm A (IC) vs Arm C (mICR); Test type: Superiority; Hazard Ratio (HR) = 0.75

2. Secondary Outcome: Proportion of Participants With an Objective Response Rate (CR or PR)
Description: Objective response is defined as either complete response or partial response. Complete response is defined as disappearance of all lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. Partial response is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Assessed every 3 months for 2 years, every 6 months for the 3rd year, then annually up to 5 years
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (IC) | Arm B (ICR) | Arm C (mICR)
Number analyzed (Participants) | 44 | 16 | 45
proportion of participants | 0.23 [0.13 to 0.35] | 0.44 [0.23 to 0.67] | 0.36 [0.24 to 0.49]
Statistical Analysis 1: Comparison: Arm A (IC) vs Arm C (mICR); Test type: Superiority; p = 0.27, Chi-squared

3. Secondary Outcome: Proportion of Patients With Grade 3 or Higher Treatment-related Adverse Events
Description: Adverse events were assessed using NCI Common Terminology Criteria for Adverse Events (CTCAE). Treatment-related adverse events are defined as those that are possibly, probably, or definitely related to protocol therapy.
Time Frame: Assessed every 2 weeks while on treatment and for 30 days after the end of treatment
Population: All patients who received protocol therapy and had toxicity data were included in this analysis.
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (IC) | Arm B (ICR) | Arm C (mICR)
Number analyzed (Participants) | 68 | 16 | 48
proportion of participants | 0.49 [0.38 to 0.59] | 0.81 [0.58 to 0.95] | 0.56 [0.43 to 0.68]

4. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from randomization to death or date last known alive.
Time Frame: Assessed every 3 months for 2 years, every 6 months for the 3rd year, then annually up to 5 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (IC) | Arm B (ICR) | Arm C (mICR)
Number analyzed (Participants) | 44 | 16 | 45
months | 19.3 [10.8 to 23.4] | 15.0 [7.06 to 22.3] | 19.2 [12.8 to 25.9]
Statistical Analysis 1: Comparison: Arm A (IC) vs Arm C (mICR); Test type: Superiority; p = 0.55, Log Rank; Hazard Ratio (HR) = 0.86

ADVERSE EVENTS:
Time Frame: Assessed every 2 weeks while on treatment and for 30 days after the end of treatment
Description: Serious adverse events are defined as grade 3 or higher adverse events that are possibly, probably, or definitely related to protocol therapy. Other adverse events are defined as grade 1 or grade 2 adverse events that are possibly, probably, or definitely related to protocol therapy with a frequency of at least 5% in a given arm.
  All patients enrolled are included in all-cause mortality analysis. Patients who received treatment with adverse event data available are included in AE analysis.
Arm/Group | Arm A (IC) | Arm B (ICR) | Arm C (mICR)
All-Cause Mortality (participants affected / at risk) | 55/70 | 15/16 | 43/50
Serious Adverse Events (participants affected / at risk) | 33/68 | 13/16 | 27/48
Other Adverse Events (participants affected / at risk) | 64/68 | 16/16 | 46/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (IC) (N=68) | Arm B (ICR) (N=16) | Arm C (mICR) (N=48)
Anemia (Blood and lymphatic system disorders) | 2 | 2 | 3
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Fatigue (General disorders) | 1 | 5 | 5
Infusion related reaction (General disorders) | 2 | 0 | 0
General and administration site - Other (General disorders) | 0 | 0 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 8 | 1 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 0
Anal mucositis (Gastrointestinal disorders) | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Colonic perforation (Gastrointestinal disorders) | 0 | 2 | 0
Diarrhea (Gastrointestinal disorders) | 8 | 3 | 7
Mucositis oral (Gastrointestinal disorders) | 1 | 2 | 3
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Rectal pain (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0
Allergic reaction (Immune system disorders) | 5 | 0 | 1
Anorectal infection (Infections and infestations) | 0 | 2 | 0
Papulopustular rash (Infections and infestations) | 1 | 0 | 0
Paronychia (Infections and infestations) | 1 | 0 | 1
Skin infection (Infections and infestations) | 1 | 0 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0
Infections and infestations - Other (Infections and infestations) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 7 | 4 | 5
Platelet count decreased (Investigations) | 0 | 1 | 2
White blood cell decreased (Investigations) | 2 | 1 | 5
Anorexia (Metabolism and nutrition disorders) | 0 | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 3 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 3 | 2 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 4 | 2 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0
Neoplasms - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Corneal ulcer (Eye disorders) | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 2
Renal and urinary disorders - Other (Renal and urinary disorders) | 0 | 0 | 1
Hematoma (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 2 | 3
Hypotension (Vascular disorders) | 2 | 0 | 0
Thromboembolic event (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (IC) (N=68) | Arm B (ICR) (N=16) | Arm C (mICR) (N=48)
Anemia (Blood and lymphatic system disorders) | 33 | 12 | 26
Chills (General disorders) | 0 | 1 | 3
Edema face (General disorders) | 0 | 1 | 1
Edema limbs (General disorders) | 6 | 3 | 7
Fatigue (General disorders) | 35 | 13 | 32
Alopecia (Skin and subcutaneous tissue disorders) | 16 | 9 | 14
Dry skin (Skin and subcutaneous tissue disorders) | 12 | 6 | 18
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Palmar-plantar erythrodysesthesia (Skin and subcutaneous tissue disorders) | 3 | 3 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 6 | 15
Rash acneiform (Skin and subcutaneous tissue disorders) | 48 | 14 | 30
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 17 | 6 | 19
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Skin and subcutaneous tissue - Other (Skin and subcutaneous tissue disorders) | 5 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 8 | 5 | 6
Anal mucositis (Gastrointestinal disorders) | 0 | 1 | 2
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 12 | 2 | 13
Diarrhea (Gastrointestinal disorders) | 36 | 12 | 30
Dry mouth (Gastrointestinal disorders) | 4 | 1 | 4
Dyspepsia (Gastrointestinal disorders) | 3 | 0 | 3
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 0 | 3
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 11 | 5 | 16
Nausea (Gastrointestinal disorders) | 29 | 11 | 20
Oral hemorrhage (Gastrointestinal disorders) | 1 | 1 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 2 | 2
Rectal pain (Gastrointestinal disorders) | 4 | 0 | 0
Stomach pain (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 18 | 6 | 10
Paronychia (Infections and infestations) | 7 | 4 | 2
Skin infection (Infections and infestations) | 0 | 1 | 0
Upper respiratory infection (Infections and infestations) | 1 | 1 | 1
Alanine aminotransferase increased (Investigations) | 10 | 4 | 8
Alkaline phosphatase increased (Investigations) | 9 | 5 | 11
Aspartate aminotransferase increased (Investigations) | 7 | 6 | 12
Lymphocyte count decreased (Investigations) | 8 | 1 | 5
Neutrophil count decreased (Investigations) | 10 | 9 | 17
Platelet count decreased (Investigations) | 17 | 8 | 20
Weight gain (Investigations) | 1 | 0 | 3
Weight loss (Investigations) | 10 | 5 | 10
White blood cell decreased (Investigations) | 25 | 11 | 21
Anorexia (Metabolism and nutrition disorders) | 15 | 8 | 16
Dehydration (Metabolism and nutrition disorders) | 4 | 2 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 3 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 | 6 | 11
Hypocalcemia (Metabolism and nutrition disorders) | 9 | 8 | 10
Hypokalemia (Metabolism and nutrition disorders) | 12 | 3 | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 28 | 9 | 26
Hyponatremia (Metabolism and nutrition disorders) | 3 | 2 | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 5
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Musculoskeletal and connective - Other (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0
Dizziness (Nervous system disorders) | 7 | 0 | 3
Dysgeusia (Nervous system disorders) | 3 | 2 | 2
Headache (Nervous system disorders) | 4 | 2 | 5
Peripheral motor neuropathy (Nervous system disorders) | 1 | 2 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 15 | 4 | 8
Blurred vision (Eye disorders) | 2 | 1 | 6
Conjunctivitis (Eye disorders) | 5 | 2 | 2
Dry eye (Eye disorders) | 1 | 2 | 5
Watering eyes (Eye disorders) | 1 | 1 | 5
Eye disorders - Other, specify (Eye disorders) | 2 | 1 | 2
Insomnia (Psychiatric disorders) | 7 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 10
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Proteinuria (Renal and urinary disorders) | 5 | 5 | 14
Hypertension (Vascular disorders) | 5 | 2 | 22
Hypotension (Vascular disorders) | 2 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-22): https://cdn.clinicaltrials.gov/large-docs/80/NCT01079780/Prot_SAP_000.pdf